CLINICAL TRIAL: NCT02816684
Title: Pegasys VR: Integrating Virtual Humans in the Treatment of Child Social Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5R42MH094019-05 (NIH)
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Anxiety Disorders
Keywords: phobic disorders; anxiety disorders
MeSH Terms: conditions — Anxiety Disorders; Phobic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SET-C (Active Comparator): Social Effectiveness Therapy for Children (SET-C; Beidel et al., 2000) includes social skills training, peer generalization experiences, and in vivo exposure.
  Interventions: Behavioral: Social Effectiveness Therapy for Children
- Pegasys-VR (Experimental): SET-C SST and individual exposure sessions are the same as the active comparator. Peer generalization sessions are replaced by a virtual environment, known as Pegasys School. children engage with artificially intelligent avatars throughout the school.
  Interventions: Behavioral: Pegasys-VR

INTERVENTIONS:
Behavioral: Pegasys-VR — Pegasys-VR uses artificially intelligent avatars and serious game technology to assist children in the acquisition and use of social skills.
  Arms: Pegasys-VR
Behavioral: Social Effectiveness Therapy for Children — Group social skills training, peer generalization sessions, individual exposure therapy
  Arms: SET-C

SUMMARY:
Among children, social anxiety is a common, severe and chronic disorder. Social Effectiveness Therapy for Children (SET-C) is an empirically supported treatment with significant potential to impact the lives of children with this severe and chronic disorder. The proposed Pegasys-VR™ system will distinctly enhance its utility, as it will allow dissemination to a broad variety of clinical settings including schools as well as traditional outpatient clinics. Its use for the treatment of social skills deficits will offer a superior solution for mental health personnel, solving many of the resource and logistic barriers that they currently face. The final product will address cost and practical issues by disseminating an empirically-supported treatment that was rigorously built and tested. Using VE will make the traditional social skills therapy programs program cost-effective and patient-centric, allowing even clinicians with little background/training in behavior therapy to have tools not typically available to them.

DETAILED DESCRIPTION:
Anxiety disorders are the most common psychiatric disorders among youth, with lifetime prevalence ranging between 18-20% of the general population. Among anxiety disorders, social anxiety disorder (SAD) affects 8% of all youth, resulting in significant short and long-term impairment, including increased likelihood of substance abuse, limited academic achievement, attenuated occupational functioning, and impaired or missing social relationships. Emerging data suggest that interventions that include social skills training, formal peer generalization sessions, and homework assignments as part of an overall treatment strategy show enhanced efficacy when compared to interventions without these components - the latter two elements which are designed to enhance skill generalization. Two critical treatment elements (peer generalization, homework assignments) are difficult to implement in traditional clinical settings, limiting optimal dissemination to youth in need of these services in different settings (e.g., at school, outpatient, or community facilities). In a recently completed Phase I STTR, the investigators developed and validated an interactive virtual environment (VE) to solve the need for intensive behavioral practice opportunities that are critical for skill generalization. The VE, known as Pegasys-VR™, allowed intensive practice of social skills without the need for formal peer group activities (in clinic solution) or intensive parental involvement (at-home solution). The results indicated that implementing a VE environment into the SET-C program was accessible, credible and feasible for the parents, clinicians and children who participated in the trial. Furthermore, examination of within group changes indicated statistically significant improvement in SAD symptoms. Given the success of the Phase I, and the need to increase the automation of the system to increase its acceptance and adoption among clinicians and socially anxiety youth, the Phase II STTR study will have the following goals: incorporate an artificial intelligence natural language system, develop additional VEs for in-clinic practice, expand the homework solution to provide additional opportunities to reinforce skills acquisition and generalization practice in in-vivo settings, using serious game theory and technology, and conduct a randomized controlled trial with youth ages 7 to 12 to test whether Pegasys-VR™ is as effective as a traditional behavioral interventions for youth with social anxiety disorder and if the effects are maintained at 3 month follow-up. If Pegasys-VR™ is clinically efficacious, it would offer a sustainable, cost-effective intervention that can be easily and rapidly disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of social anxiety disorder

Exclusion Criteria:

* an IQ < 85 and/or the presence of comorbid conduct disorder, bipolar disorder, severe depression, suicidal ideation, ADHD, developmental disorders or psychotic disorders

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Social Phobia and Anxiety Inventory for Children | Change from baseline at 12 weeks
  self-report measure of social anxiety disorder in children

SECONDARY OUTCOMES:
Diagnosis of Social Anxiety Disorder | 12 weeks
  assigned at completion of the diagnostic interview
Child Behavior Checklist | Change from baseline at 12 weeks
  parental assessment of child functioning
Child Global Assessment of Functioning | change from baseline at 12 weeks
  clinician assessment of child functioning
Clinical Global Improvement Scale | change from baseline at 12 weeks
  clinician assessment of child improvement
Behavioral Assessment | change from baseline at 12 weeks
  direct observation of child social skill

CONTACTS AND LOCATIONS:
Overall Officials: Deborah C Beidel, Ph.D., Principal Investigator — University of Central Florida
Locations (1):
- UCF RESTORES, University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No